CLINICAL TRIAL: NCT00158678
Title: Phase III Trial of Intensity-modulated Radiotherapy Plus Cisplatin Versus Conventional Radiotherapy Plus Cisplatin in Patients With Stage III-IV Head and Neck Squamous Cell Carcinoma
Brief Title: IMRT Plus Cisplatin Versus Conventional Radiotherapy Plus Cisplatin in Stage III-IV HNSCC
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2004-01
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2020-04-15 (Actual); Status verified 2020-04

CONDITIONS: Oral Cancer; Oropharynx Cancer; Hypopharynx Cancer
Keywords: oral cancer; oropharynx cancer; hypopharynx cancer; IMRT
MeSH Terms: conditions — Mouth Neoplasms; Oropharyngeal Neoplasms; Hypopharyngeal Neoplasms

ARMS (2):
- 1 (Active Comparator): Conventional RT 70Gy + concomitant cisplatin
  Interventions: Procedure: Conventional radiotherapy 70 Gy; Drug: concomitant cisplatin
- 2 (Experimental): IMRT 75Gy + concomitant cisplatin
  Interventions: Procedure: IMRT 75 Gy; Drug: concomitant cisplatin

INTERVENTIONS:
Procedure: IMRT 75 Gy — 50 Gy in PTV1 and 25 Gy in 10 fractions in PTV2
  Arms: 2
Procedure: Conventional radiotherapy 70 Gy — 50 Gy in PTV1 and 20 Gy in PTV2
  Arms: 1
Drug: concomitant cisplatin — 100 mg/m2 D1, D22, D43

SUMMARY:
This is a multicentric randomized phase III trial comparing intensity-modulated radiotherapy (75 Gy) plus cisplatin versus conventional radiotherapy (70 Gy) plus cisplatin in patients with stage III-IV squamous cell carcinoma of oral cavity, oropharynx or hypopharynx. The main end points are the rate of locoregional control and the rate of xerostomia at 2 years.

DETAILED DESCRIPTION:
This is a multicentric randomized phase III trial comparing intensity-modulated radiotherapy plus concomitant cisplatin versus conventional radiotherapy plus concomitant cisplatin in patients with stage III-IV squamous cell carcinoma of oral cavity, oropharynx or hypopharynx. The main end points are the rate of locoregional control and the rate of xerostomia at 2 years.

The IMRT total dose is 75 Gy (50 Gy to PTV1 and T0 + 25 Gy (10 fractions) to PTV2). The conventional radiotherapy total dose is 70 Gy (50 Gy to PTV1 + 20 Gy (10 fractions) to PTV2). In both arms, the cervical nodes will receive 50 Gy (65 Gy in case of Np) by conventional radiotherapy (IMRT is allowed in the IRMT arm). In the two arms, patients will receive concomitant cisplatin (100 mg/m² D1, D21, D42).

ELIGIBILITY:
Inclusion Criteria:

* squamous cell carcinoma of oral cavity, oropharynx or hypopharynx
* Stage III - IV (T1-T4, N0-N2)(UICC 2002)
* Not resected
* Indication of radiotherapy to bilateral cervical nodes at dose>= 50 Gy
* Delineation of target volumes done before randomization
* Scintigraphy of parotid gland done before radiotherapy start
* Quality of life questionnaires (EORTC-C30 and EORTC-H&N35) filled in by the patient
* Informed consent signed

Exclusion Criteria:

* N3 (UICC 2002)
* Distant metastasis
* Contra-indication to concomitant cisplatin
* History of cancer within the last 5 years
* History of head and neck radiotherapy
* Administration of drugs for treatment or prophylaxis of xerostomia (pilocarpine, ethyol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 310 (Estimated)
Dates: Start 2005-09-27 (Actual); Primary Completion 2020-03-22 (Actual); Study Completion 2020-03-22 (Actual)

PRIMARY OUTCOMES:
Loco regional control | 2 years

SECONDARY OUTCOMES:
Survival | 2 years
Xerostomia at 2 years (evaluated by parotid gland scintigraphy) | 2 years
Quality of life (EORTC-QLQ-H&N35) | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Jean Bourhis, PhD, Principal Investigator — Gustave Roussy, Cancer Campus, Grand Paris; Michel Lapeyre, MD, Principal Investigator — Centre Alexis Vautrin
Locations (2):
- France (2):
  - Centre Alexis Vautrin, Vandœuvre-lès-Nancy
  - Institut Gustave Roussy, Villejuif

REFERENCES:
- [Derived] Tao Y, Auperin A, Blanchard P, Alfonsi M, Sun XS, Rives M, Pointreau Y, Castelli J, Graff P, Wong Hee Kam S, Thariat J, Veresezan O, Heymann S, Renard-Oldrini S, Lafond C, Cornely A, Casiraghi O, Boisselier P, Lapeyre M, Biau J, Bourhis J. Concurrent cisplatin and dose escalation with intensity-modulated radiotherapy (IMRT) versus conventional radiotherapy for locally advanced head and neck squamous cell carcinomas (HNSCC): GORTEC 2004-01 randomized phase III trial. Radiother Oncol. 2020 Sep;150:18-25. doi: 10.1016/j.radonc.2020.05.021. Epub 2020 May 15. PMID 32417348